CLINICAL TRIAL: NCT05316454
Title: Effect of Self-Efficacy Support on Medication Adherence and Self-Efficacy Levels in Hypertension Patients: A Randomized Controlled Trial
Brief Title: Self-Efficacy Support on Medication Adherence and Self-Efficacy Levels in Hypertension Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bahar Ciftci, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.. 0.01.00/
Record Dates: First submitted 2022-03-21; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Hypertension
Keywords: Nursing, hypertension, self-efficacy, self-efficacy support
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients with hypertension benefit from self-efficacy support in terms of medication adherence and self-efficacy.
  Interventions: Behavioral: self-efficacy support
- Control (No Intervention): No change.

INTERVENTIONS:
Behavioral: self-efficacy support — self-efficacy support
  Arms: Experimental

SUMMARY:
Background:Health professionals are responsible for the education of hypertension patients.

Aim:The aim of this research is to see how self-efficacy support affects hypertension patients' medication adherence and self-efficacy levels.

Methods: This research is randomized controlled interventional research. The research is conducted inTurkey June-December2021.The research sample included 63hypertension patients who met the research's research requirements.According to the sequence of the arrival at the hospital, data were separated into groups with odd(intervention group)and double(control group)numbers.The necessary forms for both groups' pre-test data were filled out face-to-face. The intervention group received hands-on blood pressure measurement training with the "Hypertension Training Manual",including how to self-measure blood pressure.Over the course of the research, patients were asked to check their blood pressure twice a day at home and record the results.The patients in the intervention group were reminded of their blood pressure measurement three times a week by SMStechnique for three months to avoid forgetting it.Three months later, the same forms for the post-test data of both groups were filled out with an online survey method.The data were evaluated using the single-blind study.

DETAILED DESCRIPTION:
Background:Health professionals are responsible for the education of hypertension patients.

Aim:The aim of this research is to see how self-efficacy support affects hypertension patients' medication adherence and self-efficacy levels.

The Research's Population and Sample Hypertension patients who applied to the cardiology outpatient clinics at a Hospital in Turkey between June and December 2021 formed the target population of the research. The research sample included 63 hypertension patients over the age of 18 who met the research requirements and agreed to participate.

A priori power analysis was used to determine the sample size, and it was determined that each of the intervention and control groups needed at least 30 hypertension patients for the research's power to exceed 80% at the 95% confidence interval, 0.05 significance level, and medium effect size. Given the possibility of data loss owing to a variety of factors, it was decided to include 100 hypertension patients in the research sample. Because 12 patients wished to withdraw from the research and 25 patients did not complete the final applications, the research sample consisted of 63 hypertension patients, 31 in the intervention group and 32 in the control group.

Criteria for Research Inclusion All intervention and control groups were required to meet the inclusion criteria below.

* With a diagnosis of essential hypertension, follow up for at least 6 months,
* Using antihypertensive drugs,
* Not changing the antihypertensive medication in the last 1 month,
* Not having mental or communication problems,
* Being the age of 18 or older,
* Having at least primary education level,
* Not being a pregnant or nursing mother. Data Collection Data Collection Tools To Be Used in the Research The research data were collected using the "Patient Descriptive Information Form", "Self-Efficacy-Efficacy Scale", and "Medication Adherence Self-Efficacy-Efficacy Scale in Hypertensive Patients." Patient Introductory Information Form This form, which has been developed by the researchers based on the literature and has 19 questions, includes the socio-demographic characteristics of the patients and their disease-related features.

Self-Efficacy - Efficacy Scale The scale evaluates generic self-efficacy-efficacy perception and does not belong to any subjective category. The Self-Efficacy-Efficacy Scale is a 23-item, 5-point Likert-type scale with a minimum of 23 points and a maximum of 115 points.

Medication Adherence Self-Efficacy Scale in Hypertensive Patients The scale consists of 13 items and is in a four-point Likert type. The scale can be used to determine the lowest 13 and highest 52 points. The increase in the scale score shows that the individuals' compliance with the antihypertensive medication is above average.

Used Materials for Self-Efficacy Support Hypertension Education Booklet The Hypertension Education Booklet, which was created by the researchers based on the literature review, contains information about the disease and its treatment, treatment methods, lifestyle changes that are effective in the management of hypertension, the importance of treatment compliance, and blood pressure measurement at home.

For the booklet, 1 internal medicine specialist, 3 nurse faculty members, and 1 specialist nurse provided expert opinions. In addition, three hypertension patients were given the booklet to assess its comprehension, and arrangements were made based on their ideas. The survey was completed after Item and Content validity analyses were performed.

Blood Pressure Monitor Given the uncertainty of measurement by auscultation, the Hypertension Guidelines in the 2015 Canadian Education Program advocate using an automatic sphygmomanometer for office blood pressure measurement.Blood pressure is now measured at home using an upper arm blood pressure monitor. As a result, an appropriate blood pressure monitor, which enables self-measured blood pressure monitoring at home, with the BAP project number TSA-2021-8985 was delivered within the scope of the project. The device complies with the European Norm EN 60601-1-2.

Phone "Don't forget to measure your blood pressure in the morning and evening!" message sent 3 times a week by SMS method to the patients in the intervention group. In addition, the patients were contacted by phone at the end of the first, second, and third months to acquire information regarding the research process.

Research Implementation The objective of the research and the manner of application was explained to all patients in the intervention and control groups who met the eligibility requirements. Patients who agreed to take part in the research were required to complete an "Informed Consent Form for Volunteers." As a pre-test, both groups were given the "Patient Introductory Information Form","Self-Efficacy-Efficacy Scale", and "Medication Adherence Self-Efficacy Scale in Hypertensive Patients" through a face-to-face interview.

Separation of Groups Patients were sorted into odd and even numbers according to the order in which they arrived at the hospital in the research, regardless of their age or gender, as long as the number of participants in the intervention and control groups was equal. The method was repeated until a total of 100 data points were collected, with odd numbers representing the intervention group and even numbers representing the control group.

Intervention Group Patient education and blood pressure measurement training took place in the ECG room of the outpatient clinic which is equipped to instruct patients. The "Hypertension Education Booklet" was used to instruct the patients. Following that, the patient received blood pressure measurement training, including a demonstration of how to self-measure blood pressure. The patient was instructed to repeat the same process. The researcher provided retraining in the event of errors or shortcomings. The training continued until the patient performed the accurate measurement. It took around half an hour. The patients were given a blood pressure monitor to use at home to test their blood pressure. Patients were asked to take their blood pressure at home twice a day and record the results during the research. Patients in the intervention group were texted three times a week for three months to remind them to take their blood pressure.

The patients were called by phone after the first month to control the procedure and acquire information about the research process. In addition, the patients' queries were answered and information on the various events that occurred was acquired. Similarly, patients were also reached by phone after the second month to control the process and acquire information about the research process. The same forms were given to the patients in the intervention group as a post-test at the end of the third month, utilizing an online survey method.

Control Group The control group received no intervention after the pre-test data of the control group were gathered face to face. The same forms were collected as post-test data via an online survey method at the end of the third month.

Pre-Application The researcher invited two patients who applied to the outpatient clinic to read and answer the survey questions before the research to assess the intelligibility of the questions in the data collection form. All of the questions were found to be clear and of adequate scope. The data of the patients, taken to the pre-application, were not included in the research data.

Data Evaluation The statistics were evaluated using the single-blind study. The data were analyzed in the SPSS 20 Package Program. To establish their distribution among the groups, frequency and percentage distributions were utilized. The intervention and control groups were compared using the chi-square test. To compare two independent groups, an "independent sample t-test" was utilized. To compare two dependent groups, a "Paired t-test" was performed. Descriptive statistics (mean and standard deviation) were used. The statistical significance cut-off value was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

All intervention and control groups were required to meet the inclusion criteria below.

* With a diagnosis of essential hypertension, follow up for at least 6 months,
* Using antihypertensive drugs,
* Not changing the antihypertensive medication in the last 1 month,
* Not having mental or communication problems,
* Being the age of 18 or older,
* Having at least primary education level,
* Not being a pregnant or nursing mother.

Exclusion Criteria:

All intervention and control groups were required to meet the inclusion criteria below.

* With a diagnosis of essential hypertension, follow up for at least 6 months,
* Using antihypertensive drugs,
* Not changing the antihypertensive medication in the last 1 month,
* Not having mental or communication problems,
* Being the age of 18 or older,
* Having at least primary education level,
* Not being a pregnant or nursing mother.

Ages: 50 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy - Efficacy Scale | 3months
  The scale evaluates generic self-efficacy-efficacy perception and does not belong to any subjective category. The Self-Efficacy-Efficacy Scale is a 23-item, 5-point Likert-type scale with a minimum of 23 points and a maximum of 115 points.
Medication Adherence Self-Efficacy Scale in Hypertensive Patients | 3months
  The scale consists of 13 items and is in a four-point Likert type. The scale can be used to determine the lowest 13 and highest 52 points. The increase in the scale score shows that the individuals' compliance with the antihypertensive medication is above average.

CONTACTS AND LOCATIONS:
Overall Officials: BAHAR Çiftçi, phd, Study Director — Ataturk University
Locations (1):
- Atatürk University Faculty of Nursing, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The article is intented to be shared after it is published.

REFERENCES:
- [Derived] Erden Y, Yildiz GN, Ciftci B, Avsar G, Ozek S, Ozbek E, Sarialioglu A. The effect of self-management program with tele-nursing based on the Roper-Logan-Tierney model on self-care of hypertensive patients: a randomized controlled trial. BMC Nurs. 2025 Mar 25;24(1):313. doi: 10.1186/s12912-025-02854-y. PMID 40133854